CLINICAL TRIAL: NCT04018716
Title: Clinical Performance of MTA Cavity Lining in the Treatment of Deep Caries Lesions: A 4- Year Randomized Controlled Clinical Trial
Brief Title: Clinical Performance of MTA Cavity Lining in the Treatment of Deep Caries Lesions
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Uzay Koc, Principal Investigator, Hacettepe University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HEK 11/106
Record Dates: First submitted 2019-07-09; First posted 2019-07-12 (Actual); Last update posted 2019-07-16 (Actual); Status verified 2019-07

CONDITIONS: Mineral Trioxide Aggregate; Calcium Hydroxide; Indirect Pulp Capping
Keywords: deep dentin caries; randomized clinical trial; mineral trioxide aggregate; calcium hydroxide; total caries excavation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MTA (Experimental): mineral trioxide aggregate
  Interventions: Device: MTA
- Dycal (Active Comparator): calcium hydroxide cement
  Interventions: Device: Dycal

INTERVENTIONS:
Device: MTA — Indirect capping with MTA
  Arms: MTA
Device: Dycal — Indirect capping with Dycal
  Arms: Dycal

SUMMARY:
Aim of this clinical study is to compare the clinical success of two lining materials regarding the maintenance of pulp vitality in the treatment of deep caries lesions over 4- years.

A hundred permanent premolar and molars with deep caries lesions without pulp involvement (aged between 18 and 30 years) in 73 patients were randomly divided into the following groups: calcium hydroxide cement (Ca(OH)2) (Dycal, Dentsply/Caulk, Dentsply International Inc, Milford, DE, USA) group and mineral trioxide aggregate (MTA) (Dentsplay, Tulsa Dental, Johnson city, USA) group. Final restoration with a resin-based composite (Gradia Direct Posterior, GC, Tokyo, Japan) in a single session was performed. The following-up period was 6-, 12-, 24-, 36- and 48-months. Two calibrated examiners performed the clinical examination of the pulpal symptoms

DETAILED DESCRIPTION:
Aim of this clinical study is to compare the clinical outcomes of mineral trioxide aggregate (MTA) cavity lining with calcium hydroxide (Ca(OH)2) regarding the maintenance of pulp vitality in the treatment of deep caries lesions over 4- years.

Materials and Methods: A hundred permanent premolar and molars with deep caries lesions without pulp involvement (aged between 18 and 30 years) in 73 patients were randomly divided into the following groups: calcium hydroxide cement (Ca(OH)2) (Dycal, Dentsply/Caulk, Dentsply International Inc, Milford, DE, USA) group and mineral trioxide aggregate (MTA) (Dentsplay, Tulsa Dental, Johnson city, USA) group. Final restoration with a resin-based composite (Gradia Direct Posterior, GC, Tokyo, Japan) in a single session was performed. The following-up period was 6-, 12-, 24-, 36- and 48-months. Two calibrated examiners performed the clinical examination of the pulpal symptoms. The data will be analyzed with Pearson chi-square, Fisher exact and logrank statistics tests (p < 0.05). The Kaplan-Meier survival analysis will be conducted to reveal the survival rate.

ELIGIBILITY:
Inclusion Criteria:

1. Primary deep caries lesion with risk of pulp exposure (radiograph depth reaching 3/4 of the dentin).
2. Restorable by direct restoration and functional permanent posterior teeth,
3. Positive response to electric pulp testing and negative response to thermal testing.

Exclusion Criteria:

1. Two or more cuspal loss 2. Caries beneath the gingival margin 3. Spontaneous pain history 4. Presence of any periapical pathology 5. Immature teeth with open apex 6. Pathologic mobility

-

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 73 (Estimated)
Dates: Start 2015-07-07 (Actual); Primary Completion 2016-01-07 (Actual); Study Completion 2019-07-07 (Estimated)

PRIMARY OUTCOMES:
Evaluating of clinical success of restorations | 6 months
  The treatment consequence was judged as "clinically successful" when the following criteria were met: positive response to electric pulp testing, negative response to cold stimuli by air-water shrinkage, no general pain, normal response to tactile tests or triggered pain not lingering, no evidence of abscess, sinus tract and no abnormal tooth mobility. These teeth were considered to be "clinically healthy" and the treatment was successful.